CLINICAL TRIAL: NCT07383792
Title: From Theory to Practice: Enhancing Nurses' Clinical Skills in Bone Marrow Transplantation Through Targeted Education
Brief Title: Effect of BMT Educational Guidelines on Nurses' Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Heba Abubakr Mohamed Salama, Assistant Professor, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Bone Marrow Transplant
Record Dates: First submitted 2026-01-18; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Bone Marrow Transplantation; Nursing Performance
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nurse (Experimental): nurses caring of patients undergoing bone marrow transplantation
  Interventions: Other: education

INTERVENTIONS:
Other: education — nurse education regarding care of patients undergoing bone marrow transplantation (theoretical and practical)

SUMMARY:
implementation the educational sessions to nuses caring with BMT patients

DETAILED DESCRIPTION:
Before starting the educational guidelines, the nurses were assessed using all study tools to determine their educational needs and the number of sessions required. • Based on the findings of the assessment phase, the educational guidelines were provided to the nurses. The 'educational session' includes both a knowledge component and practical sessions. The nurses will be divided into small groups to acquire the related information.

To gather information for the observational checklist, every nurse will be observed. before and after the education in addition to knowledge assessment and attitude

ELIGIBILITY:
Inclusion Criteria:

* nurses providing direct care for adult patients undergoing bone marrow transplantation
* different qualifications
* willing to participate in the study.

Exclusion Criteria:

-

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2025-08-25 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Nurses' Knowledge Assessment Questionnaire | before education, immediately post-education, and after 3 months implementation of the targeted education
  It was designed by the researcher after reviewing relevant literature to assess nurses' practice regarding care of patients undergoing bone marrow transplantation before and after implementation of education-based guidelines. It will include the following: care of patients pre-, during, and post-bone marrow transplantation in the hospital and care after discharge from the hospital.
  Scoring system:
  Score (2) for each correct practice, (1) for needing more practice, and (zero) for not done. Total nurses' practice scores will be categorized into two levels:
  * Satisfactory ≥ 80% of total score and
  * Unsatisfactory: < 80% of total score.
Nurses' practice observational checklist | before education, immediately post-education, and after 3 months implementation of the targeted education
  It was designed by the researcher after reviewing relevant literature to assess nurses' practice regarding care of patients undergoing bone marrow transplantation before and after implementation of educational-based guidelines. It will include the following: care of patients pre-, during, and post-bone marrow transplantation in the hospital and care after discharge from the hospitals.
  Scoring system:
  Score (2) for each correct practice, (1) for needing more practice, and (zero) for not done. Total nurses' practice scores will be categorized into two levels:
  * Satisfactory ≥ 80% of total score and
  * Unsatisfactory: < 80% of total score.
Nurses Attitude Scale | before education, immediately post-education, and after 3 months implementation of the targeted education
  This scale is used to evaluate the level of nurses' attitude. It involves 15 statements aimed to assess nurses 'attitude toward stem cell therapy and the applications related to it such as stem cells collection is approved by religious, stem cells transplantation is a lifesaving treatment, and using stem cell in the trial of treatment with new drug. Attitude responses ranged from "Strongly Agree 4" "Agree3", "Disagree, 2" and" Strongly disagree, 1" for responses. The score ranged from 15 to 60, its classified into two categories: positive attitude if the score is ≥60%, and negative attitude if the score is ˂60%

CONTACTS AND LOCATIONS:
Overall Officials: Heba A Salama, Principal Investigator — Mansoura University
Locations (1):
- Faculty of Nursing, Al Mansurah, Mansoura, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol